CLINICAL TRIAL: NCT01645033
Title: Computer-based Cognitive Behavioral Therapy for Risky Behaviors in Opioid Dependent Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1111009300; P50DA009241-18 (NIH)
Record Dates: First submitted 2012-07-17; First posted 2012-07-19 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Opioid Dependence; Hepatitis; HIV
Keywords: Cognitive Behavioral Therapy; computer
MeSH Terms: conditions — Opioid-Related Disorders; Hepatitis | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAU plus computerized CBT (Experimental): Standard treatment (TAU) plus a short session using a computer program containing computerized CBT to understand risks related to sexual and other behaviors and how those risks relate to spread of infections.
  Interventions: Other: computerized Cognitive Behavioral Therapy (CBT); Other: Treatment as Usual (TAU)
- Treatment as Usual (TAU) (Active Comparator): This is the infectious disease orientation that would normally be received at this clinic to address risky behavior. This orientation generally includes individual and group therapy sessions that discuss behaviors and the resulting risk of sexually or drug-related infections (for example: use of a condom). Sessions will generally include items such as:
  * Teaching about the treatment program
  * Teaching important ideas about sexual behaviors risks
  * Increasing knowledge about specific sexually transmitted diseases
  * Discussions of ways to reduce or minimize spread of diseases related to drug use [for example, Hepatitis and Human Immunodeficiency virus (HIV, the virus responsible for causing AIDS)]
  Interventions: Other: Treatment as Usual (TAU)

INTERVENTIONS:
Other: computerized Cognitive Behavioral Therapy (CBT) — Standard treatment (as described in TAU) plus a short session using a computer program containing CBT to understand risks related to sexual and other behaviors and how those risks relate to spread of infections.
  Arms: TAU plus computerized CBT
Other: Treatment as Usual (TAU) — This is the infectious disease orientation that would normally be received at this clinic to address risky behavior. This orientation generally includes individual and group therapy sessions that discuss behaviors and the resulting risk of sexually or drug-related infections (for example: use of a condom). Sessions will generally include items such as:
  * Teaching about the treatment program
  * Teaching important ideas about sexual behaviors risks
  * Increasing knowledge about specific sexually transmitted diseases
  * Discussions of ways to reduce or minimize spread of diseases related to drug use [for example, Hepatitis and Human Immunodeficiency virus (HIV, the virus responsible for causing AIDS)]

SUMMARY:
The purpose of this study is to determine if a computerized version of Cognitive Behavioral Therapy (CBT) can improve high-risk sexual behaviors in patients attending an outpatient methadone treatment clinic. This population is at high risk for contracting and spreading hepatitis and HIV. When added to their treatment as usual (TAU), the CBT session will increase the total exposure of clients to education about how to reduce risky sexual and needle use behaviors and provides real world examples. This study seeks to determine if the use of this CBT program is easily added into the clinical program and if patients are satisfied with its use.

The main hypothesis is that the use of computerized CBT in addition to treatment as usual will improve knowledge and reduce occurrences of unprotected sexual activity. The study will also look at patient and clinic costs related to the CBT intervention, drug use and retention/adherence.

DETAILED DESCRIPTION:
We plan to conduct a randomized pilot trial evaluating the feasibility and promise of computerized CBT as a single module targeting risky sexual behavior in a HIV/Hepatitis C virus(HCV) high risk population. In the context of a drug treatment program, we will randomize 60 methadone maintenance patients to either standard treatment as usual at the program (TAU) or TAU plus the HIV/HCV/STD risk reduction module of CBT4CBT("Stay Safe"). Participants will be assessed at baseline, one month and three month time points. The primary outcome measures will be knowledge regarding risk of infection and transmission of HIV/HCV/STD,self report assessment of risky sexual practices, retention in the study and client satisfaction with the module. Our specific aims are as follows:

1. To determine the feasibility of integrating CBT4CBT/"Stay Safe" into this setting. Feasibility will be determined by completion of assessments at 1 and 3 month time points (retention) and satisfaction ratings by participants randomized to the computer module.
2. Compare knowledge of HIV/HCV/STD transmission and its prevention before and after intervention. This will be assessed by percent correct answers on a quiz administered at each assessment.
3. To evaluate changes in drug and sex risk behaviors by treatment. The primary outcome measure will be number of unprotected sexual encounters on self-assessment instruments for risky sexual behaviors.

We hypothesize that the single session of computer-based CBT will result in reduced risky sexual behaviors and increased knowledge of HIV/HCV/STD transmission with differences in retention by intervention. A successful outcome for this pilot project would result in an effect size of 0.30 or more on outcomes of risk behavior. This intervention will be compared to treatment as usual at the participating site, which currently consists of two group educational sessions on safety regarding risks of HIV/AIDS and hepatitis.

Preliminary Data- The case for computer-based behavioral treatments Computer-assisted therapies offer a relatively novel approach to the dissemination of Evidence Based Therapies (EBT) for behavioral interventions. Existing evidence points to their efficacy and cost-effectiveness. Computer-based interventions offer a number of attractive characteristics for use in primary care and substance treatment settings. Their low cost coupled with high consistency, accessibility and standardization are some associated advantages. Ease of implementation will be critical to reaching patients in remote and rural areas or in small medical offices as primary care providers become a mainstay of substance abuse treatment. Risky sexual behaviors can be targeted without the potential negative associations of face to face behavioral interventions for this highly sensitive domain and thus may be ideally modulated with computer-based therapies. Equivalency to counselor-based education for learning new health behaviors, cost-effectiveness, patient satisfaction and accessibility for illiterate patients are other advantages shown with computer-based therapy.

Computer-based CBT: Carroll et al. at Yale have developed an effective computer-based version of CBT, called "CBT4CBT" and have demonstrated its efficacy in reducing drug use and building coping skills.(38) The program makes extensive use of 'movies' as teaching tools: In each module, the user watches an individual confront a difficult situation relevant to that module's topic; after teaching the key skill through a variety of strategies, the 'movie' repeats but has a different ending because the characters implement the targeted coping skills. In developing CBT4CBT, we sought to develop an engaging version of CBT that could take advantage of the capacity of computer-based learning to convey information via a wide range of media (e.g., text, video, graphics, audio instruction, interactive exercises). The CBT4CBT program is highly user-friendly, requiring no previous experience with computers and minimal use of text-based material (i.e., minimal reading is required), and is highly interactive. In particular, we capitalize on the use of videotaped examples to allow users to actually see examples of individuals utilizing skills and strategies in a range of realistic situations. Viewers are able to watch real-life challenges acted out and safe behaviors modeled, while addressing negative or detrimental thought processes that predispose to unhealthy or risky behavior choices (e.g. making a decision to have sex without a condom). Viewer knowledge base is targeted by didactic portions and role playing is modeled by the actors. The module includes the opportunity for the client to print out and perform 'homework' worksheets, shown to be predictive for successful outcomes in CBT. The module allows for considerable control by the viewer, who can choose the speed of progression through the screens and has the capability to go back to previous screens for reviewing.

Single CBT module application: Our original feasibility, efficacy, durability and cost-effectiveness studies for addictions treatment employed the full version of CBT4CBT, comprised of 7 modules. One independent module focuses entirely on targeting risky sexual and drug use practices (titled "Stay Safe"), but has not been evaluated as an independent module for effects on risk reduction. The "Stay Safe" module was developed by Dr. Kathleen Carroll and her team at Yale in consultation with the Connecticut AIDS Education and Training Center director (Karina Danvers) and others. Its development involved the input of the CBT experts (Dr. Carroll, Dr. Michael Copenhaver), infectious disease specialists and substance abuse treatment patients who volunteered to review the module. Like the substance abuse targeted sections, the script was written to be easily recognizable across many socioeconomic and cultural groups. Professional actors were hired to play the parts of substance users in two separate high risk situations, one sexual and one Intravenous drug use (IDU). Skills are taught with multimedia presentation allowing the user to direct the pace of the module, as well as to view the consequences of various choices during the risky situation. The intervention for the proposed pilot study is this single targeted module, "Stay Safe". The module can be completed on virtually any computer, and thus is ideal for implementation in this, and a wide range of settings. Its expense for clinical use will also be reduced as a result of its brevity. These characteristics will make it easily disseminated, with "real world" applications for settings of substance use treatment and primary care medicine.

Overview: In order to maximize scientific yield from this project, we intentionally designed the study to parallel the landmark Calsyn(5) and Tross(6) randomized trials evaluating effects of the 5-session group CDC behavioral approach for risky sex practices reduction in substance abuse treatment programs. We seek to compare as closely as possible the variable of therapy type (computerized CBT in our study versus group therapy for safer sex skills building in theirs), so we sought to minimize the differences between outcome measures and methods. Use of parallels in design and outcome measures will allow us to 'benchmark' outcomes to reported changes in those studies.

Study Population and Sample: Hartford Dispensary (Hartford, CT) will serve as the site. Drug treatment and medical services are offered on an outpatient basis there. This study will enroll clients undergoing IDU treatment with methadone at the site. These clients come in regularly for scheduled maintenance medication and clinical monitoring as well as standard counseling. Many (roughly 55%) of these patients are already HCV and/or HIV positive and therefore pose a significant risk for the transmission of the virus through routes other than IDU.

Recruitment: Clients will be identified through self-presentation response to advertisements and fliers in the clinic. Drug counseling providers may also ask clients if they are interested in participating in the study. A sample size of 60 (30 patients per group) is feasible and would be sufficient to detect a large effect size on risky sexual behavior of [Cohen's d= 0.3, (alpha.05, power0.8)]. This effect size is smaller than that reported for behavioral studies in the literature, but should be sufficient to evaluate feasibility and promise of the proposed intervention in this pilot.

ELIGIBILITY:
Inclusion Criteria:

* mental capability to complete the study (as determined by MMSE, Mini Mental Status Exam score >25),
* age 18 or older,
* able to speak, read and understand English,
* actively enrolled in methadone maintenance for intravenous drug use for 30 days or longer;
* had unprotected vaginal or anal intercourse or oral sex within the past 6 months;
* not pregnant or trying to become pregnant.

Exclusion Criteria:

* have an untreated bipolar or schizophrenic disorder
* are pregnant (by self-report) or trying to become pregnant (these may unduly influence behaviors of sexual activity)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2012-04; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of unprotected sexual occurrences, measured by an assessment, the HIV Risk-taking Behavior Scale (HRBS) | 1 month (Number of unprotected sexual occurrences for the 28 days prior to completing an assessment, the HRBS)
  Self-report of unprotected sexual occurrences for the previous 28 days will be recorded; measurements are obtained at baseline, 1 month and 3 months following randomization.
Number of unprotected sexual occurrences, measured by an assessment, the HIV Risk-taking Behavior Scale (HRBS) | 3 months (Number of unprotected sexual occurrences for the 28 days prior to completing an assessment, the HRBS)
  Self-report of unprotected sexual occurrences for the previous 28 days will be recorded; measurements are obtained at baseline, 1 month and 3 months following randomization.

SECONDARY OUTCOMES:
Knowledge quiz score (measured as percent correct number of items on a knowledge quiz created for this study) | baseline (measured as percent correct number of items on a knowledge quiz created for this study)
  Knowledge on a quiz designed for this study. Answers will be true/false and % correct will be used as the outcome measure. Questions will pertain to sexual activity practices (e.g. the use of condoms), as they relate to the transmission of HCV, HIV and STD's
Knowledge quiz score (measured as percent correct number of items on a knowledge quiz created for this study) | immediately after CBT (quiz administered up to two hours following intervention), measured as percent correct number of items on a knowledge quiz created for this study
  Knowledge on a quiz designed for this study. Answers will be true/false and % correct will be used as the outcome measure. Questions will pertain to sexual activity practices (e.g. the use of condoms), as they relate to the transmission of HCV, HIV and STD's
Knowledge quiz score (measured as percent correct number of items on a knowledge quiz created for this study) | 1 month followup (measured as percent correct number of items on a knowledge quiz created for this study)
  Knowledge on a quiz designed for this study. Answers will be true/false and % correct will be used as the outcome measure. Questions will pertain to sexual activity practices (e.g. the use of condoms), as they relate to the transmission of HCV, HIV and STD's
Knowledge quiz score(measured as percent correct number of items on a knowledge quiz created for this study) | 3 month followup (measured as percent correct number of items on a knowledge quiz created for this study)
  Knowledge on a quiz designed for this study. Answers will be true/false and % correct will be used as the outcome measure. Questions will pertain to sexual activity practices (e.g. the use of condoms), as they relate to the transmission of HCV, HIV and STD's

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M Carroll, PhD, Principal Investigator — Yale University Department of Psychiatry
Locations (1):
- Hartford Dispensary, Hartford, Connecticut, United States